CLINICAL TRIAL: NCT05118581
Title: Safety and Efficacy of Ultrasound Guided Vascular Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Elsayed, resident doctor at vascular surgery department sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Soh-Med-21-10-25
Record Dates: First submitted 2021-10-13; First posted 2021-11-12 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Vascular Access; Ultrasound Guided Vascular Access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients need vascular access (Experimental): Arterial or venous cathetrization guided by ultrasound
  Interventions: Device: ultrasound guided vascular access

INTERVENTIONS:
Device: ultrasound guided vascular access — Arterial or venous catheterization guided by ultrasound

SUMMARY:
Vascular access involves central and peripheral vein accesses and arterial accesses. Central venous catheterization is widely used in clinical practice for diverse purposes, including hemodialysis for end stage renal failure, invasive hemodynamic monitoring, radiological studies, infusion of drugs that cannot be administered via peripheral vessels, administration of parenteral nutrition, vascular access in patients whose peripheral veins are difficult to be catheterized and for miscellaneous purposes that require access to large caliber vessels.

Arterial cannulation is used for invasive arterial pressure monitoring and to ensure access for diagnostic and therapeutic interventions.

In the United States and United Kingdom, guidelines have recommended the use of ultrasound guidance to reduce complications and improve success in central venous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* · Adult patients who need vascular access (arterial or venous)

Exclusion Criteria:

* · Patients with local infection in the area targeted for vascular access.

  * Patients with severe generalized infection and other skin diseases or lesions.
  * patients with history of DVT of the target vein and or pulmonary embolism.
  * Patients with untreated coagulopathy (INR >1.5 or platelets <50000mm3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse effects of ultrasound guided vascular access | one year
  Number of participants with adverse effects after ultrasound guided vascular access

IPD SHARING:
Plan to Share IPD: Undecided